CLINICAL TRIAL: NCT06340542
Title: Effectiveness of Thoracic Mobility Exercise Versus Manual Release Technique in Minimizing Mechanical Upper Back Pain Among Undergraduates in Sri Lanka
Brief Title: Comparison of Thoracic Mobility Exercise Versus Manual Release Technique in Minimizing Upper Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dhaka (Other)
Responsible Party: Principal Investigator, Vithursha Sivakumar, Principal Investigator, University of Dhaka
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDhaka
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Upper Back Pain
Keywords: Upper Back Pain; Undergraduates; Muscle strength; Thoracic Spine Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: This study is a Randomized Control Trial, Double- Blinded study. Participants and accessors was blinded. Participants were allocated randomly in to two groups which are experimental group which will receive thoracic mobility exercises and control group which will receive myofascial release and joint mobilization treatment by using lottery method.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants' allocation was concealed by using lottery method whether there are in exercise group or manual therapy group. Accessors was blinded which means they were not aware about the treatment or therapy which was obtained by the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Thoracic mobility exercises were given to the participants. Exercises has to be performed with combination of breathing which involve holding time 10 seconds 5 repetition per set, 3 sets Each exercise has to perform 5 days in a week for 2 weeks two times a day.
  Interventions: Other: Thoracic Mobility exercises
- Manual Release technique group (Active Comparator): Manual therapy including trigger point release and thoracic mobilization were applied for 3 times a week for two weeks.
  Interventions: Other: Manual Release technique

INTERVENTIONS:
Other: Thoracic Mobility exercises — Exercises which focus on improve the mobility of the spine especially thoracic region was administered to the patients in different position including quadruped and standing position.
  Arms: Exercise Group
Other: Manual Release technique — Interventions include release the muscle tension, trigger point release and reducing stiffness of spine was administered
  Arms: Manual Release technique group

SUMMARY:
Methodology: study aims to evaluate the effectiveness of thoracic mobility exercise and manual release technique in terms of pain intensity, thoracic mobility, muscle strength and improving disability.

Study Design: Study was conducted in Service unit of Department of Physiotherapy at university of peradeniya. Undergraduates who are currently having upper back pain for more than seven days was selected as sample. It is a randomized Controlled trail, Double blinded study. Participants allowed randomly to both groups which are experimental group which will receive thoracic mobility exercises and control group which will receive myofascial release and joint mobilization treatment. Total sample size was 60.

DETAILED DESCRIPTION:
Study Population: Undergraduates who are currently having upper back pain for more than seven days was selected as sample. Participants who was have sub-acute and chronic pain which means who will have pain more than a week or seven days will be selected as sample and who have subjected to any recent surgeries, recent fractures, accidents or injuries in upper back will be excluded from the study.

Study Setting:

Study was conducted in Service unit of department of Physiotherapy, University of Peradeniya.

Study Design:

This study is a Randomized Control Trial, Double- Blinded study. Participants and accessors was blinded. Participants was allocated allocated randomly in to two groups which are experimental group which receive thoracic mobility exercises and control group which will receive myofascial release and joint mobilization treatment.

Sample size was Calculated by using G*power 3.1.9.4 software by assigning power 80% effective size 0.5, type I error = 0.05 and type II error = 0.2. Therefore calculated sample size was 42. Drop down rate of participants is assigned as 25 %. Therefore final sample size which obtained was 60 (Kang, 2021). Simple Random Sampling was used as sampling technique as well as 30 Participants was randomly allocated to each group. Participant was allocated to the groups by using lottery method. Measurement tool contains two sections such as pre-test and post-test questionnaire. In Pre-test questionnaire, there are six sections which includes personal details of the participants, pain related questions, Measurement of range of motion at base line, muscle strength at base line and pain-self-efficacy Questionnaire (PSEQ) at base line.

In Post-test questionnaire, there are 4 sections which include, pain related questions mainly pain intensity after two weeks, muscle strength after two weeks, Range of motion after two weeks and pain-self-efficacy Questionnaire (PSEQ). Personal details of the participants will be collected separately for the concealed allocation and participants will be identified by code number Ethical approval will be obtained from the Institutional Review Board of Bangladesh Health Professional Institute. Written informed consent will be obtained from all the subjects who are willing to participate in the study. Participation in this research is entirely voluntary basis and the participants have the right to withdraw from the study at any time. Baseline outcome measures are demographic characteristics of participants such as age, gender, BMI, family size, bread winner of the family, monthly income and financial support for study; Pain duration; Pain intensity at present moment, sitting, forward bending, standing, walking, sleeping, transferring and pain when performing day to day activities; Range of Motion of thoraco-lumbar flexion and extension; Muscle strength of thoracic spine extensors and overall scale of Pain-Self- efficacy Questionnaire. After two weeks same outcome measures will be obtained other than demographic characteristics and pain duration Study Duration:This study will be conducted from July 2022 to July 2024, for two years with three months data collection

ELIGIBILITY:
Inclusion Criteria:

* Undergraduates who are currently having upper back pain for more than seven days will be selected as sample.
* Participants who will have sub-acute and chronic pain which means who will have pain more than a week or seven days will be selected as sample

Exclusion Criteria:

* Participant who have subjected to any recent surgeries, recent fractures, accidents or injuries in upper back will be excluded from the study.

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | at base line and after two weeks
  Visual Analogue Scale is used to measure the pain intensity in base line and after intervention in two groups in the following instances, present pain intensity and during sitting, forward bending, standing, walking, sleeping, transferring and performing day to day activities. Its 10 point grading scale, Here maximum value of the scale 10 indicates an unbearable pain and minimum value denotes no pain at all.
Range of Motion | at baseline and after two weeks
  Range of Motion of thoraco-Lumbar Flexion and Extension (Tape Measurement). Normal range of Thoraco lumbar flexion in tape measurement 2.7 cm is normal and for extension 2.5cm is normal
Muscle strength | at base line and after two week
  Muscle strength of spinal extensors examined by using Manual Muscle Test- Oxford Grading Scale. It is a 6 point grading scale which includes, 0 is considered as no contraction, 1 is palpable contraction, 2 movement with gravity eliminated, 3 is movement against gravity only, 4 movement against gravity with some resistance and 5 is movement against with full resistance
Disability level - self perception | at baseline and after two week
  Pain-Self-Efficacy-Questionnaire is used to analyse how participants feel confident despite the pain. Total score is 60. If the total score indicates more than 45 patient has a stronger self efficacy believe to the pain and if its less than 30 weak or less self efficacy believe to the pain

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Hossain, PhD, Study Chair — Head of Department of Physiotherapy, Professor of Bangladesh Health Professional Institute; Vithursha Sivakumar, B.Sc, Principal Investigator — Student of Master of Rehabilitation Science at Bangladesh Health professional Institute
Locations (1):
- Vithursha Sivakumar, Jaffna, Northern Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No
Participants demographic details such as name, contact details will be kept confidential by primary investigator until the publication. After that it will be discarded

REFERENCES:
- [Result] Felemban RA, Sofi RA, Alhebshi SA, Alharbi SG, Farsi NJ, Abduljabbar FH, Farsi JMA. Prevalence and Predictors of Musculoskeletal Pain Among Undergraduate Students at a Dental School in Saudi Arabia. Clin Cosmet Investig Dent. 2021 Feb 17;13:39-46. doi: 10.2147/CCIDE.S292970. eCollection 2021. PMID 33633467
- [Result] Lee KS, Lee JH. Effect of maitland mobilization in cervical and thoracic spine and therapeutic exercise on functional impairment in individuals with chronic neck pain. J Phys Ther Sci. 2017 Mar;29(3):531-535. doi: 10.1589/jpts.29.531. Epub 2017 Mar 22. PMID 28356648
- [Result] Kim J, Sung DJ, Lee J. Therapeutic effectiveness of instrument-assisted soft tissue mobilization for soft tissue injury: mechanisms and practical application. J Exerc Rehabil. 2017 Feb 28;13(1):12-22. doi: 10.12965/jer.1732824.412. eCollection 2017 Feb. PMID 28349028
- [Result] Niemi SM, Levoska S, Rekola KE, Keinanen-Kiukaanniemi SM. Neck and shoulder symptoms of high school students and associated psychosocial factors. J Adolesc Health. 1997 Mar;20(3):238-42. doi: 10.1016/S1054-139X(96)00219-4. PMID 9069025

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT06340542/Prot_SAP_ICF_000.pdf